CLINICAL TRIAL: NCT05768126
Title: Prediction of ECT Treatment Response and Reduction of Cognitive Side-effects Using EEG and Rivastigmine
Acronym: PRECISER
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); St. Antonius Hospital (Other); Tergooi Hospital (Other)
Responsible Party: Principal Investigator, Iris Sommer, Professor, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 202000842
Record Dates: First submitted 2021-08-26; First posted 2023-03-14 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Depressive Disorder
Keywords: electroconvulsive therapy; rivastigmine; EEG
MeSH Terms: conditions — Depressive Disorder | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rivastigmine (Experimental): Rivastigmine, transdermal administration with a dosage of 4.6 and 9.6mg. The patches will be administered daily. The duration will equate to the duration of ECT treatment (that will be clinically determined)
  Interventions: Drug: Rivastigmine Transdermal Product
- Sham (Sham Comparator): Non-active patches will be administered daily. The duration will equate to the duration of ECT treatment (that will be clinically determined)
  Interventions: Other: Sham

INTERVENTIONS:
Drug: Rivastigmine Transdermal Product — The patches will be administered (first four weeks 4.6 mg and then 9.5. mg).
  Arms: Rivastigmine
Other: Sham — The sham patches will be administered during the same period of time as the rivastigmine.
  Arms: Sham

SUMMARY:
The goal of this clinical trial is to test the beneficial effects of rivastigmine administration, and predict the treatment outcome with electroencephalography (EEG), in patients with severe depression treated with electroconvulsive therapy (ECT). The study has two main objectives:

* to study whether rivastigmine would ameliorate the side-effect profile of ECT
* to develop an outcome prediction model based on resting state EEG for both the response to treatment as well as its side effect

Participants will be assessed by:

* Cognitive tests
* Questionnaires of clinical symptoms
* Questionnaires of depressive symptoms
* Bloodsample
* Resting state and task-based EEG

Researchers will compare patients with a depressive disorder treated with ECT receiving rivastigmine to placebo patches to see if rivastigmine reduces cognitive side effects.

DETAILED DESCRIPTION:
Electroconvulsive therapy (ECT) is the most potent psychiatric treatment, with an effect size of 1.5 for severe and refractory unipolar and bipolar depression. ECT convincingly outperforms pharmacotherapy such as tricyclic antidepressants and monoamine oxidase inhibitors and any form of psychotherapy. Despite its outstanding performance in reducing depressive symptoms up to the point of full remission, it is used only marginally. One reason for its infrequent use may be that the response to ECT is largely unpredictable, while cognitive side-effects occur frequently.

In a previous study, the researchers found that multiple cognitive tests showed a significant decline immediately post-ECT, which resolved within 6 months after the last ECT session without further treatment. Even though cognitive side-effects are mostly short-lasting, both patients and doctors see this as a great drawback of ECT. If these disturbing side-effects could be prevented, more patients and psychiatrists would choose ECT as a treatment option. This would lead to a more effective treatment and hence shorter duration of chronic severe depression and improvement in quality of life, while costs for health care and loss of productivity would decrease. A potential way of ameliorating side effects, could be to add a cholinesterase inhibitor to ECT treatment. Rodent studies show that the loss of cholinergic fibers specifically correlated to the cognitive side effects of rodents after electroconvulsive stimulation (ECS). The researchers selected rivastigmine (a cholinesterase inhibitor) as a potential candidate in counteracting cognitive side effects induced by cholinergic fiber loss due to ECT. Rivastigmine patches are very well tolerated and widely used for Alzheimer's and Parkinson's dementia.

Tailoring treatment to patients that are likely to respond while cognitive side-effects are unlikely to occur, would be another important improvement for depressed patients. Currently, ECT outcome is unpredictable. Factors that favor response include older age, psychotic depression, shorter duration of the depressive episode, and smaller volumes of the dentate gyrus (a part of the hippocampus). However, these predictors do not provide enough accuracy to make individual response profiles. Accurately classifying specifically non-responders will prevent application of ineffective treatment with potential iatrogenic damage, while more accurately predicted response will increase the applicability of ECT as treatment option. A potentially powerful way that is easy to implement in the clinic is prediction of ECT response using resting state EEG characteristics in addition to clinical information.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Clinical indication for ECT (as indicated by the treating physician/psychiatrist)
* Uni- or bipolar depression (as assessed by the treating psychiatrist)
* Fluent in Dutch

Exclusion Criteria:

* Currently receiving, or having received ECT 6 months prior to the start of the treatment/study.
* Currently using rivastigmine, galantamine, donepezil (all cholinesterase inhibitors for mild to moderate Alzheimer's Disease).
* Pregnancy and/or lactation/breast feeding
* Suspicion of neurodegenerative disorders (as diagnosed earlier)
* Contraindications for ECT (recent myocardial infarction, recent cerebrovascular accident, recent intracranial surgery, pheochromocytoma and instable angina pectoris)
* Contraindications for rivastigmine (bradycardia or atrioventricular (AV) conduction disorders (first degree AV-block excluded)
* Patients who have had an allergic reaction to rivastigmine
* Cognitive disorder not explained by the depressive episode

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-29 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
The effect of rivastigmine on scores of the verbal fluency test. | Baseline, within 72 hours after the first treatment session, within 1 week after the last treatment session and at 3-months after the last treatment session
  Changes in cognitive functioning as measured by scores on the Verbal fluency test, in which participants are asked to pronounce as many words (0 - infinity) as possible in 60 seconds in a certain category or starting with a certain letter. A higher score means a better outcome.
The effect of rivastigmine on scores of the Rey auditory verbal learning test | Baseline, within 72 hours after the first treatment session, within 1 week after the last treatment session and at 3-months after the last treatment session
  Changes in cognitive functioning as measured by scores on the Rey auditory verbal learning test, in which the assessor reads a list of of 15 words to the participant, and the participant is asked to repeat as many words as they remember. This is repeated 5 times (learning) and 15 minutes later the participant is asked how many words (0-15 words) they remember (memory). The scale ranges from 0-90 words in total. A higher score means a better outcome.
The effect of rivastigmine on changes in scores on the Montreal Cognitive Assessment | Baseline, within 72 hours after the first treatment session, within 1 week after the last treatment session and at 3-months after the last treatment session
  Changes in cognitive functioning as measured by scores on the Montreal Cognitive Assessment, that comprises of assessing multiple cognitive domains with a scoring scale of 0-30. A higher score means a better outcome.
The effect of rivastigmine on changes in scores on the Columbia University Autobiographical Memory Interview short form | Baseline, within 72 hours after the first treatment session, within 1 week after the last treatment session and at 3-months after the last treatment session
  Changes in cognitive functioning before, during and after treatment as measured by scores on the Columbia University Autobiographical Memory Interviewshort form. The subject's ability to remember the specific details originally provided during the pre-treatment interview is measured on a scale of 0-60 points. A higher score means a better outcome.
Changes in resting-state EEG peak frequency | Baseline, within 72 hours after the first treatment session, within 1 week after the last treatment session and at 3-months after the last treatment session
  To develop an outcome prediction model the investigators will use resting state EEG output in units of peak frequency
Treatment response | Baseline
  Treatment response defined as 50% symptom reduction as measured with the Hamilton Depression Scale (17-item version), that comprises of 17 questions on depressive symptoms measured on a scale of 0-52 points. A higher score means a worse outcome.
Treatment response | Within 72 hours after the first treatment session
  Treatment response defined as 50% symptom reduction as measured with the Hamilton Depression Scale (17-item version), that comprises of 17 questions on depressive symptoms measured on a scale of 0-52 points. A higher score means a worse outcome.
Treatment response | Within 1 week after the last treatment session
  Treatment response defined as 50% symptom reduction as measured with the Hamilton Depression Scale (17-item version), that comprises of 17 questions on depressive symptoms measured on a scale of 0-52 points. A higher score means a worse outcome.
Treatment response | At 3-months after the last treatment session
  Treatment response defined as 50% symptom reduction as measured with the Hamilton Depression Scale (17-item version), that comprises of 17 questions on depressive symptoms measured on a scale of 0-52 points. A higher score means a worse outcome.
Remission | Baseline
  with the Hamilton Depression Scale (17-item version), that comprises of 17 questions on depressive symptoms measured on a scale of 0-52 points. A higher score means a worse outcome. Remission as measured by a score of <7.
Remission | Within 72 hours after the first treatment session
  with the Hamilton Depression Scale (17-item version), that comprises of 17 questions on depressive symptoms measured on a scale of 0-52 points. A higher score means a worse outcome. Remission as measured by a score of <7.
Remission | Within 1 week after the last treatment session
  with the Hamilton Depression Scale (17-item version), that comprises of 17 questions on depressive symptoms measured on a scale of 0-52 points. A higher score means a worse outcome. Remission as measured by a score of <7.
Remission | At 3-months after the last treatment session
  with the Hamilton Depression Scale (17-item version), that comprises of 17 questions on depressive symptoms measured on a scale of 0-52 points. A higher score means a worse outcome.Remission as measured by a score of <7.

SECONDARY OUTCOMES:
Quality of life of patients assessed with the European Quality of Life Five Dimensions with Five Levels (Euro-QoL-5D-5L) | Baseline, within 72 hours after the first treatment session, within 1 week after the last treatment session and at 3-months after the last treatment session
  The assessment of the quality of life of patients during the study, it comprises of 5 questions, measured on a scale of 5-25. A higher score means a worse outcome.
Quality of life of patients assessed with the visual analog scale of the European Quality of Life Five Dimensions with Five Levels (Euro-QoL-5D-5L) | Baseline, within 72 hours after the first treatment session, within 1 week after the last treatment session and at 3-months after the last treatment session
  The assessment of the quality of life of patients during the study. The instrument includes a visual analog scale (VAS) anchored by 0 (worst imaginable health) and 100 (best imaginable health). A higher score means a better outcome.
Changes in the global assessment of disability using the World Health Organization Disability Assessment Schedule (WHODAS) 2.0 12 item version | Baseline, within 72 hours after the first treatment session, within 1 week after the last treatment session and at 3-months after the last treatment session
  The assessment of global disability of the patients during the study, measured on a scale of 12-60. A higher score means a worse outcome.
Changes in peak amplitude measured with selective attention EEG task | Baseline, within 72 hours after the first treatment session, within 1 week after the last treatment session and at 3-months after the last treatment session
  The selective attention tasks measures behavioral outcomes by hits/misses/false alarms.
Changes in behavioral outcome measured with the selective attention EEG task | Baseline, within 72 hours after the first treatment session, within 1 week after the last treatment session and at 3-months after the last treatment session
  The selective attention task measures behavioral outcomes by hits/misses/false alarms.
Changes in processing negativity measured with the selective attention EEG task | Baseline, within 72 hours after the first treatment session, within 1 week after the last treatment session and at 3-months after the last treatment session
  The selective attention task measures behavioral outcomes by hits/misses/false alarms.
Changes in mismatch negativity measures (amplitude, latency and duration) obtained with the MisMatch Negativity Paradigm during an EEG recoding | Baseline, within 72 hours after the first treatment session, within 1 week after the last treatment session and at 3-months after the last treatment session
  The mismatch negativity task measures event-related potentials by EEG and the Mismatch Negativity Paradigm
Change in subjective feeling of memory impairment on the Subjective Assessment of Memory Impairment (SAMI) questionnaire | Baseline, within 72 hours after the first treatment session, within 1 week after the last treatment session and at 3-months after the last treatment session
  The Subjective Assessment of Memory Impairment is a questionnaire that comprises of two questions of which the first question concerns the subjective feeling of memory point, rated on a 10-point likert scale, and is rated from 0 no impairment, to 10 severe impairment. A higher score means a worse outcome.
Change in impact of cognitive adverse events on the Subjective Assessment of Memory Impairment (SAMI) questionnaire | Baseline, within 72 hours after the first treatment session, within 1 week after the last treatment session and at 3-months after the last treatment session
  The Subjective Assessment of Memory Impairment is a questionnaire that comprises of two questions of which the second question concerns the impact of cognitive adverse events, on a 5-point likert scale, rated from 1 no complaints, to 5 severe complaints. A higher score means a worse outcome.
Changes in the Expectation of response form | Baseline, within 72 hours after the first treatment session, within 1 week after the last treatment session and at 3-months after the last treatment session
  The likelihood that they will recover questioned by a scale with a range from -5 (negative effect expected) to 5 (positive effect expected)

OTHER OUTCOMES:
Changes in Free speech using the PRAAT task | Baseline, within 72 hours after the first treatment session, within 1 week after the last treatment session and at 3-months after the last treatment session
  The researchers will collect free speech data (5 minutes of free speech) to study language characteristics of responders (remitters) and non-responders (non-remitters).
Changes in DNA methylation | Baseline, within 72 hours after the first treatment session, within 1 week after the last treatment session and at 3-months after the last treatment session
  The researchers will collect 6ml blood samples for DNA methylation levels

CONTACTS AND LOCATIONS:
Overall Officials: Iris EC Sommer, PhD, MD, Principal Investigator — UMC Groningen
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No